CLINICAL TRIAL: NCT05607823
Title: Adding Core Stabilization Training to Orofacial Manuel Therapy in Individuals With Temporomandibular Joint Disc Displacement With Reduction: A Randomized Controlled Study
Brief Title: Adding Core Stabilization Training to Manuel Therapy in Temporomandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2022.951
Record Dates: First submitted 2022-10-22; First posted 2022-11-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2022-10

CONDITIONS: Temporomandibular Joint Disorders
Keywords: core stability; exercise; Temporomandibular joint disorders; facial pain; comprehensive health care
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity; Facial Pain

STUDY DESIGN:
Intervention Model Description: There are three study groups: 1.CST group: Participants in this group will be received core stabilization training, orofacial manuel therapy and conventional physiotherapy (Home exercise program and patient education). 2. OMT group: Participants in this group will be received orofacial manuel therapy and conventional physiotherapy (Home exercise program and patient education) as treatment. 3. Control Group: Participants in this group received only conventional physiotherapy (Home exercise program and patient education) as treatment.
Who Masked: Participant
Masking Description: Participants did not know which treatment group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CST Group (Experimental): The core stabilization group. Participants in this group will be received core stabilization training, orofacial manuel therapy and conventional physiotherapy (Home exercise program and patient education) as treatment. The number of participants is planned to be 15.
  Interventions: Other: Core Stabilization Training; Other: Orofacial Manual Therapy; Other: Conventional Physiotherapy
- OMT Group (Experimental): The orofacial manuel therapy group. Participants in this group will be received orofacial manuel therapy and conventional physiotherapy (Home exercise program and patient education) as treatment. The number of participants is planned to be 15.
  Interventions: Other: Orofacial Manual Therapy; Other: Conventional Physiotherapy
- Control Group (Experimental): Participants in this group will be received only conventional physiotherapy (Home exercise program and patient education) as treatment. The number of participants is planned to be 15.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Core Stabilization Training — Core Stabilization training will be based on dynamic neuromuscular stabilization and consists of three stages. In the first session, it is to teach the simultaneous activation of the transversus abdominis, pelvic floor, multifidus and diaphragm muscles and to improve muscle coordination and proprioception in the entire spinal region. In the second and third phases, exercises will be made more intense to improve muscular endurance and stability. The difficulty of the exercises will be increased by working in different positions, using resistance bands, exercise balls and body weight, and adding movements to the extremities. A total of 10 sessions of treatment program will be applied to the patients for ten weeks, once a week.
  Arms: CST Group
Other: Orofacial Manual Therapy — As orofacial manual therapy, soft tissue (intraoral and extraoral trigger point therapy and myofascial release of painful muscles) and joint mobilization (caudal and ventro-caudal traction, ventral and mediolateral translation), muscle energy technique, fascia mandibularis release, occipital release and ligamentous treatment was planned.
  Arms: CST Group; OMT Group
Other: Conventional Physiotherapy — Conventional physiotherapy consists of home exercise and patient education. Patient education consists of parafunctional behaviors, habits, a diet with soft food, and posture education. The exercises consist of exercises for the mandible, cervical and thoracic region and breathing. All movements are planned to be done at home 3 times a day, every day of the week.

SUMMARY:
This study aims to compare the effectiveness of three different treatment approaches in individuals with DDwR symptoms. It is hypothesized that adding core stabilization training (CST) to orofacial manual therapy (OMT) will enhance treatment outcomes. Patients will be treated for 10 sessions once a week, for a total of 10 weeks. Evaluation was planned to be done twice, at the beginning and end of the treatment.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of three different treatment approaches in individuals with DDwR symptoms. It is hypothesized that adding core stabilization training (CST) to orofacial manual therapy (OMT) will enhance treatment outcomes. The patients to be included in the study will be randomly divided into three groups and it is planned to include 15 people in each group. Home exercises and patient education will be provided to all patients.

* Group 1 (CST group): Orofacial manual therapy + core stabilization training (CST) + home exercise and patient education
* Group 2 (OMT group): Orofacial manual therapy (OMT) + home exercise and patient education
* Group 3 (Control group): Home exercise and patient education.

Pain intensity, pressure pain threshold, joint range of motion, posture, flexibility, stabilization of core muscles, functionality and sleep quality will be evaluated by using Numeric Pain Scale (NPS), digital algometer, ruler, Palpation Meter (PALM), bubble inclinometer, tape measure, Finger-to-floor distance (EPZM) and sit-reach test, pressure biofeedback unit, "Helkimo Index", "Pittsburgh Sleep Quality Index (PUKI)" respectively. Patients will be treated for 10 sessions once a week, for a total of 10 weeks. Evaluation was planned to be done twice, at the beginning and end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate,
* Aged between 18-60 years old,
* Having the diagnosis of Temporomandibular Disorders (TMD) - Reduction Disc Displacement (DDwR)

Exclusion Criteria:

* Having a malignant condition, trauma and surgery of the cranial and cervical region,
* Not being cooperative,
* Regular use of analgesic and anti-inflammatory drugs,
* Having dentofacial anomalies,
* Having active arthritis,
* Having lumbal pathology,
* Having metabolic diseases,
* Having connective tissue, rheumatological and hematological disorders,
* Having a diagnosed psychiatric illness,
* Receiving TMD-related physical therapy less than 6 months ago

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Pain severity: VAS | Change from Baseline pain severity at 10 weeks.
  The severity of pain in the orofacial region was evaluated using a Numeric Pain Scale (NPS). The patients were instructed to mark the level of pain felt during rest, clenching and maximum mouth opening on a 10-cm line ranging from 0 (no pain) to 10 (intolerable pain).
Pain Threshold: Digital algometer | Change from Baseline pain threshold at 10 weeks.
  The algometer is a reliable instrument for measuring the sensitivity of the masticatory muscles. The measurement will be made at 8 points. A force (Newton in force) of 1 kg (weight in kilogram) per square centimeter (surface area in centimeter square) is applied to the patient for 3 seconds, and this is continued until the patient feels pain (weight and surface area will be combined to report Newton in kg/ cm2). The physiotherapist will passively support the individual's head with the other hand. This process will be repeated three times and the average value will be calculated.
Range of Motion | Change from Baseline range of motion at 10 weeks.
  Mouth opening, protrusion and right and left lateral deviation will be measured starting from 0 using a 15 cm ruler. Repeated measuring reduces the standard error of measurement, hence repeated measurements were also included in our study (three times) with the largest recorded range taken.
Facial asymmetry | Change from Baseline facial asymmetry at 10 weeks.
  For facial asymmetry evaluation, the distance between the anterior notch of the chin and the mandible line will be measured with a tape measure.
Degree of pelvic tilt | Change from Baseline degree of pelvic tilt at 10 weeks.
  Palpation Meter (PALM), (Salt Lake City, United Kingdom, USA) will be used for pelvic tilt evaluation. The Palpation Meter has an angle inclinometer and two 360-swivel arms, one of arms will be placed in the Spina iliaca Anterior Superior (SIAS) and the other in the Spina iliaca Posterior Superior (SIPS). In this position, the angle indicated by the inclinometer will be recorded as the pelvic tilt angle.
Degree of lordosis | Change from Baseline degree of lordosis at 10 weeks.
  Bubble inclinometer (White Plains, New York 10602 USA) will be used for lumbar lordosis evaluation. The degree of lordosis will be determined by measuring the spinous processes of the T12-L1 and S2-3 vertebrae with a bubble inclinometer and adding the degrees found.

SECONDARY OUTCOMES:
Flexibility of lumbal extensor muscles | Change from Baseline Finger-to-floor distance (EPZM) at 10 weeks.
  Finger-to-floor distance (EPZM) will be used for flexibility of lumbal extensor. In the EPZM test, individuals will stand on a stool and are asked to bend their torso forward to reach as far as possible with both hands without bending the knees. The distance between the stool level and the middle finger will be measured by the therapist and and this distance will be recorded in cm. The individual will be asked to repeat this movement three times and the highest value will be taken as the test score.
Flexibility of hamstring muscles | Change from Baseline sit-reach test at 10 weeks.
  Sit-reach test will be used for flexibility of hamstring muscles. For the sit-and-reach test, the individual will be seated without shoes in a long sitting position on the floor, with his feet propped on a 30 cm bench that is scaled by dividing the top into cm. The body will be asked to lie forward on the coffee table as much as possible without bending the knees, wait 2 seconds at the extreme point where the fingers are extended, and this distance will be recorded in cm. The individual will be asked to repeat this movement three times and the highest value will be taken as the test score.
Performance of stabilizer muscles | Change from Baseline lumbopelvic stabilization at 10 weeks.
  Lumbopelvic stabilization will be assessed using a pressure biofeedback unit (Stabilizer Pressure Biofeedback Unit, Chattanooga Group Inc., Hixson, Tennessee, USA). Individuals will be asked to lie on their back in a hooked position. The pressure cell of the instrument will be placed under the lumbar vertebrae. The subjects will be asked to perform the abdominal drawing-in maneuver as previously taught, with no spinal or pelvic movement. The change in pressure will be recorded in mmHg and the time that the contraction can be maintained in seconds.
Functionality | Change from Baseline Helkimo Index at 10 weeks.
  "Helkimo Index" will be used to evaluate Temporomandibular Joint (TMJ) pain and dysfunction. This index evaluates the clinical dysfunction of the stomatognathic system based on the 5 signs of TMD. Pain during mandible movement, TMJ pain, pain in masticatory muscles, TMJ sound and maximum mouth opening are evaluated with different questions between 0-5. The total dysfunction score ranges from 0 to 25. 0 no dysfunction; Values 1-4 are mild dysfunction; Values from 4 to 9 indicate moderate dysfunction; Values above 9 indicate severe dysfunction.
Sleep | Change from Baseline Pittsburgh Sleep Quality Index (PUKI) at 10 weeks.
  "Pittsburgh Sleep Quality Index (PUKI)" will be used to assess sleep quality and impairment. It consists of 7 subscales that assess subjective sleep quality, sleep latency and duration, habitual sleep efficiency, sleep disorders, use of sleep medication, and loss of daytime functionality. A high total score indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Kuru Colak, Asst. Prof, Study Director — Marmara University Institute of Health Sciences
Locations (1):
- Sultan İğrek, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study.

REFERENCES:
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Liu F, Steinkeler A. Epidemiology, diagnosis, and treatment of temporomandibular disorders. Dent Clin North Am. 2013 Jul;57(3):465-79. doi: 10.1016/j.cden.2013.04.006. PMID 23809304
- [Background] Anastassaki Kohler A, Hugoson A, Magnusson T. Prevalence of symptoms indicative of temporomandibular disorders in adults: cross-sectional epidemiological investigations covering two decades. Acta Odontol Scand. 2012 May;70(3):213-23. doi: 10.3109/00016357.2011.634832. Epub 2011 Nov 30. PMID 22126531
- [Background] Nekora-Azak A, Evlioglu G, Ordulu M, Issever H. Prevalence of symptoms associated with temporomandibular disorders in a Turkish population. J Oral Rehabil. 2006 Feb;33(2):81-4. doi: 10.1111/j.1365-2842.2006.01543.x. PMID 16457666
- [Background] Hoffmann RG, Kotchen JM, Kotchen TA, Cowley T, Dasgupta M, Cowley AW Jr. Temporomandibular disorders and associated clinical comorbidities. Clin J Pain. 2011 Mar-Apr;27(3):268-74. doi: 10.1097/AJP.0b013e31820215f5. PMID 21178593
- [Background] Lee KC, Wu YT, Chien WC, Chung CH, Chen LC, Shieh YS. The prevalence of first-onset temporomandibular disorder in low back pain and associated risk factors: A nationwide population-based cohort study with a 15-year follow-up. Medicine (Baltimore). 2020 Jan;99(3):e18686. doi: 10.1097/MD.0000000000018686. PMID 32011444
- [Background] Cuccia A, Caradonna C. The relationship between the stomatognathic system and body posture. Clinics (Sao Paulo). 2009;64(1):61-6. doi: 10.1590/s1807-59322009000100011. PMID 19142553
- [Background] Gangloff P, Louis JP, Perrin PP. Dental occlusion modifies gaze and posture stabilization in human subjects. Neurosci Lett. 2000 Nov 3;293(3):203-6. doi: 10.1016/s0304-3940(00)01528-7. PMID 11036196
- [Background] Espinosa de Santillana IA, Garcia-Juarez A, Rebollo-Vazquez J, Ustaran-Aquino AK. [Frequent postural alterations in patients with different types of temporomandibular disorders]. Rev Salud Publica (Bogota). 2018 May-Jun;20(3):384-389. doi: 10.15446/rsap.V20n3.53529. Spanish. PMID 30844014
- [Background] Saito ET, Akashi PM, Sacco Ide C. Global body posture evaluation in patients with temporomandibular joint disorder. Clinics (Sao Paulo). 2009;64(1):35-9. doi: 10.1590/s1807-59322009000100007. PMID 19142549
- [Background] Fischer MJ, Riedlinger K, Gutenbrunner C, Bernateck M. Influence of the temporomandibular joint on range of motion of the hip joint in patients with complex regional pain syndrome. J Manipulative Physiol Ther. 2009 Jun;32(5):364-71. doi: 10.1016/j.jmpt.2009.04.003. PMID 19539119
- [Background] Fink M, Wahling K, Stiesch-Scholz M, Tschernitschek H. The functional relationship between the craniomandibular system, cervical spine, and the sacroiliac joint: a preliminary investigation. Cranio. 2003 Jul;21(3):202-8. doi: 10.1080/08869634.2003.11746252. PMID 12889677
- [Background] de Oliveira-Souza AIS, de O Ferro JK, Barros MMMB, Oliveira DA. Cervical musculoskeletal disorders in patients with temporomandibular dysfunction: A systematic review and meta-analysis. J Bodyw Mov Ther. 2020 Oct;24(4):84-101. doi: 10.1016/j.jbmt.2020.05.001. Epub 2020 May 11. PMID 33218570
- [Background] von Piekartz H, Hall T. Orofacial manual therapy improves cervical movement impairment associated with headache and features of temporomandibular dysfunction: a randomized controlled trial. Man Ther. 2013 Aug;18(4):345-50. doi: 10.1016/j.math.2012.12.005. Epub 2013 Feb 14. PMID 23415640
- [Background] Wright EF, Domenech MA, Fischer JR Jr. Usefulness of posture training for patients with temporomandibular disorders. J Am Dent Assoc. 2000 Feb;131(2):202-10. doi: 10.14219/jada.archive.2000.0148. PMID 10680388
- [Background] Kalamir A, Pollard H, Vitiello A, Bonello R. Intra-oral myofascial therapy for chronic myogenous temporomandibular disorders: a randomized, controlled pilot study. J Man Manip Ther. 2010 Sep;18(3):139-46. doi: 10.1179/106698110X12640740712374. PMID 21886424
- [Background] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Background] Urbanski P, Trybulec B, Pihut M. The Application of Manual Techniques in Masticatory Muscles Relaxation as Adjunctive Therapy in the Treatment of Temporomandibular Joint Disorders. Int J Environ Res Public Health. 2021 Dec 8;18(24):12970. doi: 10.3390/ijerph182412970. PMID 34948580
- [Background] von Piekartz H, Ludtke K. Effect of treatment of temporomandibular disorders (TMD) in patients with cervicogenic headache: a single-blind, randomized controlled study. Cranio. 2011 Jan;29(1):43-56. doi: 10.1179/crn.2011.008. PMID 21370769
- [Background] Frank C, Kobesova A, Kolar P. Dynamic neuromuscular stabilization & sports rehabilitation. Int J Sports Phys Ther. 2013 Feb;8(1):62-73. PMID 23439921
- [Background] Walker N, Bohannon RW, Cameron D. Discriminant validity of temporomandibular joint range of motion measurements obtained with a ruler. J Orthop Sports Phys Ther. 2000 Aug;30(8):484-92. doi: 10.2519/jospt.2000.30.8.484. PMID 10949505
- [Background] Tuzun C, Yorulmaz I, Cindas A, Vatan S. Low back pain and posture. Clin Rheumatol. 1999;18(4):308-12. doi: 10.1007/s100670050107. PMID 10468171
- [Background] Herrington L. Assessment of the degree of pelvic tilt within a normal asymptomatic population. Man Ther. 2011 Dec;16(6):646-8. doi: 10.1016/j.math.2011.04.006. Epub 2011 Jun 11. PMID 21658988
- [Background] Perret C, Poiraudeau S, Fermanian J, Colau MM, Benhamou MA, Revel M. Validity, reliability, and responsiveness of the fingertip-to-floor test. Arch Phys Med Rehabil. 2001 Nov;82(11):1566-70. doi: 10.1053/apmr.2001.26064. PMID 11689977
- [Background] Mayorga-Vega D, Merino-Marban R, Viciana J. Criterion-Related Validity of Sit-and-Reach Tests for Estimating Hamstring and Lumbar Extensibility: a Meta-Analysis. J Sports Sci Med. 2014 Jan 20;13(1):1-14. eCollection 2014 Jan. PMID 24570599
- [Background] Richardson CA, Jull GA. Muscle control-pain control. What exercises would you prescribe? Man Ther. 1995 Nov;1(1):2-10. doi: 10.1054/math.1995.0243. PMID 11327788
- [Background] Hodges P, Richardson C, Jull G. Evaluation of the relationship between laboratory and clinical tests of transversus abdominis function. Physiother Res Int. 1996;1(1):30-40. doi: 10.1002/pri.45. PMID 9238721
- [Background] Helkimo M. Studies on function and dysfunction of the masticatory system. II. Index for anamnestic and clinical dysfunction and occlusal state. Sven Tandlak Tidskr. 1974 Mar;67(2):101-21. No abstract available. PMID 4524733
- [Background] Thilander B, Rubio G, Pena L, de Mayorga C. Prevalence of temporomandibular dysfunction and its association with malocclusion in children and adolescents: an epidemiologic study related to specified stages of dental development. Angle Orthod. 2002 Apr;72(2):146-54. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 11999938
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Tuncer AB, Ergun N, Tuncer AH, Karahan S. Effectiveness of manual therapy and home physical therapy in patients with temporomandibular disorders: A randomized controlled trial. J Bodyw Mov Ther. 2013 Jul;17(3):302-8. doi: 10.1016/j.jbmt.2012.10.006. Epub 2012 Nov 16. PMID 23768273
- See also: Investigation of the Relationship Between Temporomandibular Disorder and Postural Analysis. — https://clinicaltrials.gov/ct2/show/NCT03490643
- See also: Assessment of Temporomandibular Joint Dysfunctions and the Position of Pelvis — https://www.jotsrr.org/abstract/assessment-of-temporomandibular-joint-dysfunctions-and-the-position-of-pelvis-2269.html
- See also: Manual Therapy for Temporomandibular Disorders: A Review of the Literature. J Body Mov Ther. — https://www.semanticscholar.org/paper/Manual-therapy-for-temporomandibular-disorders%3A-A-Kalamir-Pollard/eff17b74aec032c4f05e66879a61cd158ddda70d
- See also: Effects of Core Stability Exercises, Lumbar Lordosis and Low- Back Pain: A Systematic Review. — https://www.semanticscholar.org/paper/Effects-of-Core-Stability-Exercises%2C-Lumbar-and-A-%C5%A0kundri%C4%87-Vuki%C4%87evi%C4%87/47619c8a9f55f65a910228f96be0b0debffebcc6
- See also: Pressure pain threshold and pain perception in temporomandibular disorder patients: is there any correlation? — https://www.scielo.br/j/rdor/a/dV5P7vngMkggzjZqKrCvHsR/?lang=en
- See also: The Validity and Reliability of the Pittsburgh Sleep Quality Index — https://www.turkpsikiyatri.com/turkceOzet?Id=327